CLINICAL TRIAL: NCT01619696
Title: Prospective Pilot Study of Multimodal Radiological Evaluation Feasibility During Chemoradiotherapy of Rectal Adenocarcinomas.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0932103
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Rectal Adenocarcinoma
Keywords: chemotherapy; rectal adenocarcinoma; proctectomy; Fmiso TEP; MRI
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Procedure: Pelvic MRI and F MISO TEP

INTERVENTIONS:
Procedure: Pelvic MRI and F MISO TEP — Pelvic MRI and F MISO TEP: before inclusion, 2 weeks after beginning and 7 weeks after completion of chemoradiotherapy.

SUMMARY:
The objective of the present project is to validate the feasibility of a multimodal radiological pathway while on chemoradiotherapy, in order to validate potentially predictive factors for chemoradiotherapy sensitivity of rectal adenocarcinomas.

DETAILED DESCRIPTION:
The objective of the present project is to validate the feasibility of a multimodal radiological pathway while on chemoradiotherapy, in order to validate potentially predictive factors for chemoradiotherapy sensitivity of rectal adenocarcinomas.

It is based on a structured clinical and radiological pathway for patients, using diffusion MRI and F misonidazole PET.

Validation of these new tools is already needed in clinical practice since future institutional trials will be based on treatment individualisation, using preoperative predicting factors.

ELIGIBILITY:
Inclusion Criteria:

* locally advanced (≥T3) resectable rectal adenocarcinoma between 2 and 10 cm from the anal verge.

Exclusion Criteria:

* synchonous metastatis
* previous malignant tumour
* previous radiotherapy/ chemotherapy
* performance status WHO>2
* contraindication to 5 FU

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
acceptation rate of the entire sequence by eligible patients | 13 weeks
  acceptation rate of the entire sequence by eligible patients

SECONDARY OUTCOMES:
radiological changes while on chimiotherapy, to tumour regression, and prognosis | 13 weeks
  radiological changes while on chimiotherapy, to tumour regression, and prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Portier, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, Toulouse, France